CLINICAL TRIAL: NCT06050343
Title: Comparative Study of the Pharmacokinetics and Pharmacodynamics of Rinsulin® R, Solution for Injection, 100 IU/ml (GEROPHARM LLC) and Humulin® Regular, Solution for Injection, 100 IU/ml (Eli Lilly) in Euglycemic Hyperinsulinemic Clamp Method
Brief Title: Comparative Study of Rinsulin R (GEROPHARM) and Humulin Regular (Eli Lilly) Euglycemic Hyperinsulinemic Clamp Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RINCL-R
Record Dates: First submitted 2020-08-03; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Bioequivalence; Therapeutic Equivalency
Keywords: human recombinant insulin; euglycemic hyperinsulinemic clamp
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Crossover Assignment two-way crossover
Who Masked: Participant, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rinsulin® R (Experimental): Single subcutaneous administration of Insulin at a dose 0.3 IU / kg
  Interventions: Drug: Humulin® Regular; Drug: Rinsulin® R
- Humulin® Regular (Active Comparator): Single subcutaneous administration of Insulin at a dose 0.3 IU / kg
  Interventions: Drug: Humulin® Regular; Drug: Rinsulin® R

INTERVENTIONS:
Drug: Humulin® Regular — subcutaneous injection at a dose of 0.3 IU / kg
  Other Names: Reference drug
Drug: Rinsulin® R — subcutaneous injection at a dose of 0.3 IU / kg
  Other Names: Test Drug

SUMMARY:
Pharmacokinetics and pharmacodynamics of Rinsulin® R, injection solution, 100 IU / ml (GEROPHARM LLC, Russia) and Humulin® Regular, injection solution, 100 IU / ml (Lilly France ", France) using the euglycemic hyperinsulinemic clamp method.

DETAILED DESCRIPTION:
A double-blind, randomized, comparative, crossover study of the pharmacokinetics and pharmacodynamics of Rinsulin® R, solution for injection, 100 IU / ml (GEROPHARM LLC, Russia) and Humulin® Regular, solution for injection, 100 IU / ml (Lilly France, France) using euglycemic hyperinsulinemic clamp method on healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Men of the Caucasian race with a verified diagnosis "healthy" according to the data of standard clinical, laboratory and instrumental examination methods.
* Age 18-50, inclusive.
* Body mass index 18.5 - 27 kg / m2.
* Volunteers who have sexual contact with fertile women should agree to use barrier methods of contraception while participating in the study (unless they have undergone surgical sterilization). Study Participants must also not become a sperm donor within the specified period.
* Consent to all restrictions imposed during the study.

Exclusion Criteria:

* Acute inflammatory diseases within 3 weeks from the moment of complete recovery to the stage of screening.
* Presence of episodes of hypoglycemia in the history of the volunteer
* Presence in the family history of the closest relatives cases of verified diagnosis of diabetes mellitus of any type.
* Deviations from the norm of basic vital indicators (heart rate, blood pressure, respiratory rate, body temperature) and ECG from normal values and laboratory values from reference values during screening.
* Fasting plasma glucose> 6.1 mmol / L at screening.
* HbA1C> 6% at the time of screening.
* Oral glucose tolerance test - blood glucose level ≥7.8 mmol / L (2 hours after glucose loading) during screening.
* Hard-to-reach veins of the upper extremities, vein thrombosis, history of thrombophlebitis or family history of close relatives, "compromised" veins due to frequent preceding venipuncture.
* Taking medications, phytopreparations, biologically active additives within 14 days before screening.
* Significant blood loss 3 months before screening due to, for example, but not limited to the following points: a. donor blood donation; b. extended surgery or trauma leading to significant blood loss.
* Incomplete recovery from surgery or surgery scheduled while the volunteer is participating in the study.
* Mental, physical and other reasons interferes with adequately assessing behavior and correctly fulfill the conditions of the research protocol (incl. a history of mental illness).
* Presence or history (three years before the the study drug) of narcotic, drug and / or substance abuse.
* Positive test for the content of narcotic drugs in urine during the screening period.
* Anamnestic information about alcoholism or taking more than 10 units. alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of dry wine or 50 ml of spirits).
* Positive test for alcohol in breath during screening.
* Nicotine addiction (regular use of tobacco less than 6 months before screening).
* Any chronic diseases, incl. but not limited to positive test results for hepatitis C or hepatitis B, HIV, syphilis at the time of screening.
* Burdened allergological history.
* Presence of suspicion of an inflammatory disease of the urinary system based on the results of urinalysis during screening.
* Presence of oncological diseases within 5 years before the screening.
* History of organ transplantation (except of corneal transplant performed more than 3 months before the first injection of the study drug).
* Participation in a clinical trial of any drug or experimental medical device within 3 months prior to the first administration of the study drug.
* Any other condition that, in the reasonable opinion of the research physician, makes it difficult for the volunteer to participate in the study.

History of hypersensitivity to heparin, insulin or any of the excipients of the investigational drugs.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Смах | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Drug Observed Maximum Plasma Concentration
AUC 0-10 | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 10 h
AUC GIR 0-12 | - 120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 12 h
GIRmax | -120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Time to reach maximum glucose infusion rate

SECONDARY OUTCOMES:
tGIRmax | -120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Time to reach maximum glucose infusion rate
AUC 0-2 | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 2 h
AUC 0-4 | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 4 h
AUC 0-6 | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Total area under the curve "drug concentration - time" in the time interval from 0 to 6 h
Tmax | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Time to reach test drug Maximum Plasma Concentration
T1/2 | -60 minutes, -30 minutes, 0, every 15 minutes till 4 hours and then every 30 minutes till 10 hours
  Half-life of a test drug
tGIRlag | -120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Time between the drug administration and the onset of action
AUC GIR 0-2 | -120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 2 h
AUC GIR 0-4 | - 120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 4 h
AUC GIR 0-6 | -120 minutes, -90 minutes, -60 minutes, -30 minutes, 0, every 5 minutes till 8 hours, then every 10 minutes till 10 hours and then every 30 minutes till 12 hours
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 6 h

CONTACTS AND LOCATIONS:
Locations (1):
- "National Medical Research Center of Endocrinology" of the Ministry of Health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No